CLINICAL TRIAL: NCT00381043
Title: Campral (Acamprosate) Treatment of Alcohol Dependence in a Family Medicine Setting: A Randomized, Double-Blind Placebo-Controlled Study
Brief Title: Study of Campral (Acamprosate) for Alcohol Dependence in a Family Medicine Clinic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Wisconsin, Milwaukee (Other)
Responsible Party: Principal Investigator, James Garbutt, MD, Professor of Psychiatry, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CMP-MD-06
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Results first posted 2013-03-22 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Alcohol Dependence
Keywords: Alcohol Dependence; Family Medicine Setting; University of North Carolina at Chapel Hill
MeSH Terms: conditions — Alcoholism | interventions — Acamprosate; Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1- Acamprosate (Active Comparator): The study is a double-blind, randomized, placebo-controlled clinical trial in which participants will receive 333 mg t.i.d. oral acamprosate or matching placebo for a 12-week period. Each participant will also receive brief behavioral intervention at each visit.
  Interventions: Drug: Acamprosate (Campral)
- 2 - Sugar Pill - Placebo (Placebo Comparator): The study is a double-blind, randomized, placebo-controlled clinical trial in which participants will receive 333 mg t.i.d. oral acamprosate or matching placebo for a 12-week period. Each participant will also receive brief behavioral intervention at each visit.
  Interventions: Drug: Acamprosate (Campral)

INTERVENTIONS:
Drug: Acamprosate (Campral) — The study is a double-blind, randomized, placebo-controlled clinical trial in which participants will receive 333 mg t.i.d. oral acamprosate or matching placebo for a 12-week period. Each participant will also receive brief behavioral intervention at each visit.
  Other Names: Acamprosate, campral, alcohol dependence medication

SUMMARY:
This is a study of a medication, acamprosate, which is an FDA approved medication for alcohol problems. We will be examining whether acamprosate compared to a sugar pill (placebo) is more effective for helping with drinking in a Family Medicine clinic.

DETAILED DESCRIPTION:
Acamprosate has been shown to reduce drinking days in alcohol dependent patients and promote abstinence, with few reported side effects. A limitation of these studies, however, has been their lack of generalizability due to restrictive inclusion and exclusion criteria. Furthermore, most of the previous studies of acamprosate have been conducted in Europe, in a different treatment setting from the typical American Family Medicine center, where alcohol dependent patients are most likely to be first identified in the U.S.

The present study is designed to determine the efficacy of acamprosatefor alcohol dependence in a Family Medicine setting using minimal psychotherapeutic interventions-as would also likely occur in a primary care setting. The study will be a 12-week, double-blind, placebo-controlled, randomized trial comparing 666 mg acamprosate t.i.d. to placebo in patients at the UNC Family Medicine Center with alcohol dependence. Subjects will be seen by Family Medicine physicians and receive brief motivational interventions. Primary efficacy will be determined by measuring % days abstinent and secondary outcomes include rates of complete abstinence, % heavy drinking days, CGI and GGT in the acamprosate group compared to the placebo group.

ELIGIBILITY:
INCLUSION CRITERIA:

* 1. Men and women ages 21 to 65 years with a diagnosis of alcohol dependence.
* 2. History of at least 2 heavy drinking days (men > 5 drinks/day; women > 4 drinks/day) per week, on average, during the month prior to screening.
* 3. Ability to understand and sign written informed consent.
* 4. Willingness to refrain from drinking for at least three days prior to randomization.
* 5. Willingness to consider a goal of abstinence or a significant reduction in drinking as an objective.

EXCLUSION CRITERIA:

* 1. Clinically significant medical disease that might interfere with the evaluation of the study medication or present a safety concern.
* 2. Clinically significant psychiatric disease, e.g. bipolar disorder, psychosis, that might interfere with study participation or present a safety concern. [Subjects with depression or an anxiety disorder who are receiving medication and are clinically stable for at least one month will not be excluded.]
* 3. Suicidal ideation or behavior, history of suicide attempt.
* 4. Renal Impairment; estimated creatinine clearance <50 ml/min.
* 5. Substance use disorder other than alcohol or nicotine dependence or cannabis abuse.
* 6. Pregnant or breastfeeding women and women of childbearing potential who do not practice a medically acceptable form of birth control (oral or depot contraceptive, or barrier methods such as diaphragm or condom with spermicidal).
* 7. Individuals requiring inpatient treatment or more intense outpatient treatment for their alcohol dependence. Individuals may be considered for the trial upon completion of medical detoxification.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JC Garbutt, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - UNC Family Medicine Center, Chapel Hill, North Carolina
  - Center for Addiction and Behavioral Health Research University of Wisconsin-Milwaukee, Milwaukee, Wisconsin

REFERENCES:
- [Background] Paille FM, Guelfi JD, Perkins AC, Royer RJ, Steru L, Parot P. Double-blind randomized multicentre trial of acamprosate in maintaining abstinence from alcohol. Alcohol Alcohol. 1995 Mar;30(2):239-47. PMID 7662044
- [Background] Pelc I, Verbanck P, Le Bon O, Gavrilovic M, Lion K, Lehert P. Efficacy and safety of acamprosate in the treatment of detoxified alcohol-dependent patients. A 90-day placebo-controlled dose-finding study. Br J Psychiatry. 1997 Jul;171:73-7. doi: 10.1192/bjp.171.1.73. PMID 9328500
- [Background] Sass H, Soyka M, Mann K, Zieglgansberger W. Relapse prevention by acamprosate. Results from a placebo-controlled study on alcohol dependence. Arch Gen Psychiatry. 1996 Aug;53(8):673-80. doi: 10.1001/archpsyc.1996.01830080023006. PMID 8694680
- [Derived] Berger L, Fisher M, Brondino M, Bohn M, Gwyther R, Longo L, Beier N, Ford A, Greco J, Garbutt JC. Efficacy of acamprosate for alcohol dependence in a family medicine setting in the United States: a randomized, double-blind, placebo-controlled study. Alcohol Clin Exp Res. 2013 Apr;37(4):668-74. doi: 10.1111/acer.12010. Epub 2012 Nov 7. PMID 23134193

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1- Acamprosate | 2 - Sugar Pill - Placebo
Started | 51 | 49
Completed | 39 | 41
Not Completed | 12 | 8
Not completed — Lost to Follow-up | 8 | 6
Not completed — Withdrawal by Subject | 3 | 1
Not completed — wanted more care | 0 | 1
Not completed — incarcerated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1- Acamprosate | 2 - Sugar Pill - Placebo | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (7.7) | 47.7 (8.5) | 47.1 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 38
  Male | 30 | 32 | 62
Region of Enrollment [Number; unit: participants]
  United States | 51 | 49 | 100

OUTCOME MEASURES:

1. Secondary Outcome: Retention
Description: Number of individuals retained in the trial by acamprosate vs placebo group
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | 1- Acamprosate | 2 - Sugar Pill - Placebo
Number analyzed (Participants) | 51 | 49
participants | 39 | 41

2. Primary Outcome: % Dropout
Description: Percentage of participants who dropped out of study by drug condition
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | 1- Acamprosate | 2 - Sugar Pill - Placebo
Number analyzed (Participants) | 51 | 49
percentage of participants | 21.5 | 16.3

3. Primary Outcome: Percent Days Abstinent
Description: %Days without any alcohol consumption over the treatment period
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | 1- Acamprosate | 2 - Sugar Pill - Placebo
Number analyzed (Participants) | 51 | 49
percentage of days | 40.7 (30.6) | 41.6 (33.0)

4. Secondary Outcome: Percent With Complete Abstinence
Description: % of subjects with no drinking during the 12 week treatment trial
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | 1- Acamprosate | 2 - Sugar Pill - Placebo
Number analyzed (Participants) | 51 | 49
percentage of participants | 5.9 | 19.1

5. Secondary Outcome: % Heavy Drinking Days During Trial
Description: % of Heavy drinking days (5 or more drinks/d for a man or 4 or more drinks/d for a woman) over the 12 weeks of the trial.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of heavy drinking days
Arm/Group | 1- Acamprosate | 2 - Sugar Pill - Placebo
Number analyzed (Participants) | 51 | 49
percentage of heavy drinking days | 15.8 (21.3) | 18.4 (23.4)

6. Secondary Outcome: Clinical Global Impression Scale
Description: Range of overall severity of illness: 1, normal, not at all ill; 2, borderline ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1- Acamprosate | 2 - Sugar Pill - Placebo
Number analyzed (Participants) | 51 | 49
units on a scale | 2.3 (0.9) | 2.4 (1.2)

7. Secondary Outcome: % Compliant With Medication
Description: % of individuals with evidence for 80% compliance with medication based on returned blister packs and weekly diaries.
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | 1- Acamprosate | 2 - Sugar Pill - Placebo
Number analyzed (Participants) | 51 | 49
percentage of participants | 93.3 | 91.6

ADVERSE EVENTS:
Arm/Group | 1- Acamprosate | 2 - Sugar Pill - Placebo
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/49
Other Adverse Events (participants affected / at risk) | 17/51 | 12/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1- Acamprosate (N=51) | 2 - Sugar Pill - Placebo (N=49)
Diarrhea (Gastrointestinal disorders) | 17 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less